CLINICAL TRIAL: NCT05843279
Title: Efficacy of a Physiotherapy Treatment in Newborns With Breastfeeding Difficulties
Brief Title: Physiotherapy in the Treatment of Breastfeeding Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Gemma María López Segura, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35/2022
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Breastfeeding; Ankyloglossia; Lactation Disorders
Keywords: Breastfeeding; Ankyloglossia; Physiotherapy; Myofunctional Therapy; breastfeeding session
MeSH Terms: conditions — Breast Feeding; Ankyloglossia; Lactation Disorders | interventions — Myofunctional Therapy

STUDY DESIGN:
Intervention Model Description: Myofunctional Therapy is performed in one group and a breastfeeding session is performed in another group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A physiotherapist outside the study was in charge of carrying out the first evaluation in the first week of life of the infant. Another physiotherapist was in charge of applying the physiotherapy intervention. After completion of the intervention, all infants were reassessed by another physiotherapist outside the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofunctional therapy (Experimental): The intervention group receives myofunctional therapy sessions in which orofacial exercises are performed.
  Interventions: Procedure: Myofunctional therapy
- Breastfeeding session (Other): In this group, a session is held in which the posture and attachment of the baby to the mother's chest is assessed and corrected.
  Interventions: Procedure: Myofunctional therapy

INTERVENTIONS:
Procedure: Myofunctional therapy — In one group, physiotherapy intervention is performed on the orofacial structures of the baby and in another group, the posture presented by the mother while breastfeeding her baby is corrected.
  Other Names: Breastfeeding session

SUMMARY:
The objective of this randomized, single-blind clinical trial is to compare the efficacy of two treatments (Myofunctional Therapy and breastfeeding sessions) in infants who have difficulty breastfeeding during the first week of life.

The main questions to be answered are:

* Is breastfeeding improved with this type of intervention?
* What type of intervention is better?
* After carrying out these interventions, does the baby need to undergo surgery if it presents a sublingual frenulum? Participants must be infants who are one week old and who have been diagnosed with ankyloglossia through the Hazelbaker Scale. They will be randomly distributed into the two intervention groups and after one month of treatment, they will be assessed again using the same scale.

The researchers will compare the results between these two groups in order to verify the best intervention.

DETAILED DESCRIPTION:
Infants who met the inclusion and exclusion criteria, respectively, were accepted to participate in the study. The randomization of the sample was performed by a statistician, who had no prior contact with either the infants or the parents. The online Randomizer (www.randomizer.org) program was used to randomly generate 200 sets of numbers, each containing two numbers ranging from 1 to 2 in random order. After signing the consent, a code was randomly chosen for each patient, thus ensuring that the 200 patients were equally distributed into two groups according to the group number of each code: group 1 (Myofunctional Therapy group) and group 2 (group sessions lactation).

Infants who met the inclusion criteria were referred to the rehabilitation and physiotherapy service. A physical therapist outside the study was in charge of evaluating the measurements of all infants during the first week of life through all the scales detailed below (pre-test). After randomly assigning the infants, another physiotherapist was responsible for applying the intervention once a week for 30 minutes for a period of 30 days. Once the intervention was finished, all the infants (both intervention groups) were reassessed by the physiotherapist outside the study using the same baseline scales (post-test).

ELIGIBILITY:
Inclusion Criteria:

* Full-term infants exclusively breastfed
* Born both by normal delivery and by cesarean section
* Who presented difficulty in breastfeeding

Exclusion Criteria:

* Preterm newborns
* With low birth weight (less than 2,500 kg)
* Mothers with flat or inverted nipples
* Patients who did not wish and did not authorize to participate in the study.

Ages: 7 Days to 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Hazelbaker scale | one month
  This scale evaluates the appearance (5 items) and the function of the language (7 items). Each item is scored on a 2/1/0 scale (2 equals good appearance and/or full function; 1 equals moderate appearance and/or partial function; 0 equals no appearance and inadequate function). The maximum appearance score is 10, indicating that there are no limitations in the orofacial structures, and if it is less than 8, a limitation is confirmed. The maximum function score is 14, which reflects preserved function and if it is less than 11, the function is considered to be diminished.
Latch Scale | one month
  It is made up of different areas of assessment: how the baby latches on, amount of audible swallowing, type/condition of the mother's nipple, mother's comfort level, and amount of help the mother needs to latch on. baby at the breast The rating system is 0/1/2 in each item (0 equals the "least favourable" and 2 the "most favourable"). The highest score is 10, which means that there is no problem in breastfeeding. If the score is less than 9, it means that the mother and baby need help with breastfeeding.

SECONDARY OUTCOMES:
Visual Analogue Scale | one month
  This scale evaluates the pain suffered by the mother's nipple while the child is breastfeeding. The maximum score is 10 (unbearable pain) and the minimum score is 0 (no pain). Higher scores mean more breastfeeding problems and the need for help from a health professional.
Surgical intervention after treatment | one month
  If the baby needs frenectomy or frenotomy after the month of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Raúl Romero Del Rey, Almería, Almeria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messner AH, Walsh J, Rosenfeld RM, Schwartz SR, Ishman SL, Baldassari C, Brietzke SE, Darrow DH, Goldstein N, Levi J, Meyer AK, Parikh S, Simons JP, Wohl DL, Lambie E, Satterfield L. Clinical Consensus Statement: Ankyloglossia in Children. Otolaryngol Head Neck Surg. 2020 May;162(5):597-611. doi: 10.1177/0194599820915457. Epub 2020 Apr 14. PMID 32283998
- [Background] Frenectomy for the Correction of Ankyloglossia: A Review of Clinical Effectiveness and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2016 Jun 15. Available from http://www.ncbi.nlm.nih.gov/books/NBK373454/ PMID 27403491
- [Background] Ghaheri BA, Cole M, Fausel SC, Chuop M, Mace JC. Breastfeeding improvement following tongue-tie and lip-tie release: A prospective cohort study. Laryngoscope. 2017 May;127(5):1217-1223. doi: 10.1002/lary.26306. Epub 2016 Sep 19. PMID 27641715
- [Background] Bruney TL, Scime NV, Madubueze A, Chaput KH. Systematic review of the evidence for resolution of common breastfeeding problems-Ankyloglossia (Tongue Tie). Acta Paediatr. 2022 May;111(5):940-947. doi: 10.1111/apa.16289. Epub 2022 Feb 21. PMID 35150472
- [Background] Walker RD, Messing S, Rosen-Carole C, McKenna Benoit M. Defining Tip-Frenulum Length for Ankyloglossia and Its Impact on Breastfeeding: A Prospective Cohort Study. Breastfeed Med. 2018 Apr;13(3):204-210. doi: 10.1089/bfm.2017.0116. Epub 2018 Mar 20. PMID 29620937
- [Background] Ballard JL, Auer CE, Khoury JC. Ankyloglossia: assessment, incidence, and effect of frenuloplasty on the breastfeeding dyad. Pediatrics. 2002 Nov;110(5):e63. doi: 10.1542/peds.110.5.e63. PMID 12415069
- [Result] Campanha SMA, Martinelli RLC, Palhares DB. Association between ankyloglossia and breastfeeding. Codas. 2019 Feb 25;31(1):e20170264. doi: 10.1590/2317-1782/20182018264. PMID 30810632
- [Result] Colombari GC, Mariusso MR, Ercolin LT, Mazzoleni S, Stellini E, Ludovichetti FS. Relationship between Breastfeeding Difficulties, Ankyloglossia, and Frenotomy: A Literature Review. J Contemp Dent Pract. 2021 Apr 1;22(4):452-461. PMID 34267016
- [Result] Costa-Romero M, Espinola-Docio B, Paricio-Talayero JM, Diaz-Gomez NM. Ankyloglossia in breastfeeding infants. An update. Arch Argent Pediatr. 2021 Dec;119(6):e600-e609. doi: 10.5546/aap.2021.eng.e600. English, Spanish. PMID 34813240
- [Result] Brzecka D, Garbacz M, Mical M, Zych B, Lewandowski B. Diagnosis, classification and management of ankyloglossia including its influence on breastfeeding. Dev Period Med. 2019;23(1):79-87. doi: 10.34763/devperiodmed.20192301.7985. PMID 30954985
- [Result] Wen Z, Walner DL, Popova Y, Walner EG. Tongue-tie and breastfeeding. Int J Pediatr Otorhinolaryngol. 2022 Sep;160:111242. doi: 10.1016/j.ijporl.2022.111242. Epub 2022 Jul 20. PMID 35930834
- [Result] Manipon C. Ankyloglossia and the Breastfeeding Infant: Assessment and Intervention. Adv Neonatal Care. 2016 Apr;16(2):108-13. doi: 10.1097/ANC.0000000000000252. PMID 27003478
- [Result] Gonzalez Garrido MDP, Garcia-Munoz C, Rodriguez-Huguet M, Martin-Vega FJ, Gonzalez-Medina G, Vinolo-Gil MJ. Effectiveness of Myofunctional Therapy in Ankyloglossia: A Systematic Review. Int J Environ Res Public Health. 2022 Sep 28;19(19):12347. doi: 10.3390/ijerph191912347. PMID 36231647
- [Result] Ferres-Amat E, Pastor-Vera T, Rodriguez-Alessi P, Ferres-Amat E, Mareque-Bueno J, Ferres-Padro E. The prevalence of ankyloglossia in 302 newborns with breastfeeding problems and sucking difficulties in Barcelona: a descriptive study. Eur J Paediatr Dent. 2017 Dec;18(4):319-325. doi: 10.23804/ejpd.2017.18.04.10. PMID 29380619
- [Result] Ferres-Amat E, Pastor-Vera T, Rodriguez-Alessi P, Ferres-Amat E, Mareque-Bueno J, Ferres-Padro E. Management of Ankyloglossia and Breastfeeding Difficulties in the Newborn: Breastfeeding Sessions, Myofunctional Therapy, and Frenotomy. Case Rep Pediatr. 2016;2016:3010594. doi: 10.1155/2016/3010594. Epub 2016 Aug 30. PMID 27688921
- See also: Recommendations on the duration of breastfeeding according to the World Health Organization (OMS) — https://www.who.int/es/